CLINICAL TRIAL: NCT00938756
Title: Interest of the Dosage of CA 15-3 in CSF for Diagnosing Carcinomatous Meningitis in Breast Cancer
Brief Title: Study of Cerebrospinal Fluid Samples in Diagnosing Carcinomatous Meningitis in Patients With Cancer or Meningeal Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Oscar Lambret (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000633542; COL-MENINCA; COL-IDRCB-2008-A00185-50; COL-0801; INCA-RECF0807
Record Dates: First submitted 2009-07-11; First posted 2009-07-14 (Estimated); Last update posted 2010-04-07 (Estimated); Status verified 2010-04

CONDITIONS: Brain and Central Nervous System Tumors; Breast Cancer; Metastatic Cancer
Keywords: leptomeningeal metastases; male breast cancer; stage IV breast cancer; tumors metastatic to brain; adult meningioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Breast Neoplasms; Neoplasm Metastasis; Meningeal Carcinomatosis; Breast Neoplasms, Male; Brain Neoplasms; Meningioma | interventions — Immunoenzyme Techniques; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Other: diagnostic laboratory biomarker analysis
Other: immunoenzyme technique
Procedure: magnetic resonance imaging

SUMMARY:
RATIONALE: Studying samples of cerebrospinal fluid from patients with cancer or meningeal syndrome may help doctors identify biomarkers related to cancer.

PURPOSE: This clinical trial is studying cerebrospinal fluid samples in diagnosing carcinomatous meningitis in patients with cancer or meningeal syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the validity of determining CA 15-3 levels in the cerebrospinal fluid (CSF) using automated immuno-enzymatic methods.

Secondary

* Determine the sensitivity and specificity of these assays in assessing CA 15-3 in CSF.
* Assess favorability of intrathecal production of CA 15-3.
* Determine threshold interpretations of CA 15-3 levels in CSF.

OUTLINE: This is a multicenter study.

Within 15 days of suspected meningeal involvement, blood and cerebrospinal fluid samples are collected. Samples are examined by immunoenzyme assays. Patients with suspected cases of carcinomatous meningitis undergo cerebrospinal MRI.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosis of metastatic breast cancer with evidence suggestive of carcinomatous meningitis, with or without brain metastasis
  * Other type of cancer with evidence suggestive of carcinomatous meningitis
  * Meningeal syndrome without context of cancer

PATIENT CHARACTERISTICS:

* No other prior cancers
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* No prior intrathecal treatment
* At least 4 weeks since prior interferon
* No concurrent participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
CA 15-3 levels in cerebrospinal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Le Rhun, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France